CLINICAL TRIAL: NCT01375790
Title: Neuromuscular Training With Whole Body Vibration in Older People: A Randomized Multicentre Clinical Trial With Blinded to Evaluator
Brief Title: Whole-body Vibration Training in Older People
Acronym: GERIAPLAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asociacion Colaboracion Cochrane Iberoamericana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GERIAPLAT/1; PI/180-2010 (Other Grant/Funding Number: IMSERSO)
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Aging
Keywords: whole-body vibration; older people; exercise; body balance; muscle performance; falls; physiotherapy
MeSH Terms: conditions — Motor Activity | interventions — Exercise Therapy; Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise with Whole-body vibration platform (Experimental): Exercise with Whole-body vibration (WBV) platform (Power Plate®). The participants will perform static/dynamic exercises (balance and resistance training) on a vibratory platform (Frequency: 30-35 Hz; Amplitude: 2-4 mm). Training volume and intensity we will increase systematically over six weeks according to the overload principle.
  Interventions: Device: Exercise with Whole-body vibration platform
- Exercise (Active Comparator): The participants will perform the same static/dynamic exercises (balance and resistance training) like WBV group but without the vibration stimuli, during a six weeks training period (3sessions/week). Training volume and intensity we will increase systematically over six weeks according to the overload principle
  Interventions: Other: Exercise

INTERVENTIONS:
Device: Exercise with Whole-body vibration platform — The participants will perform static/dynamic exercises (balance and resistance training) on a vibratory platform (Frequency: 30-35 Hz; Amplitude: 2-4 mm).
  Other Names: Power Plate® Whole-body vibration platform
  Arms: Exercise with Whole-body vibration platform
Other: Exercise — The participants will perform the same static/dynamic exercises (balance and resistance training) like WBV group but without the vibration stimuli.
  Other Names: Balance and resistance training
  Arms: Exercise

SUMMARY:
This is a randomized, multicentre, and parallel clinical trial with blinded to evaluator.

The principal hypothesis is that whole-body vibration training plus exercise improves the body balance and prevents falls more than only exercise training in institutionalized older people. The number needed of patients is 160 (80 per group).

ELIGIBILITY:
Inclusion Criteria:

* Institutionalized older people who were 65 years and older
* The patient consent to participate in the study

Exclusion Criteria:

* Residents who present an acute disease that not resolved during 10 days.
* Residents with a pacemaker (or serious cardiac alterations)
* Residents with epilepsy
* Residents with a high risk of thromboembolism
* Residents with a history of a hip or knee joint replacement
* Residents who not were musculoskeletal disorders and cognitive or physical dysfunction that interfering with test and training procedures.
* Residents that not accept to participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Body balance. | at 6 weeks
  Body balance will be evaluated using Tinetti Test, and Timed up and go test

SECONDARY OUTCOMES:
Body balance | at six months
  Body balance will be evaluated using Tinetti Test, and Timed up and go test
Muscle performance | at 6 weeks, and 6 months
  It will be evaluated by five-sit-to-stand test, and Smartcoach Encoder.
Number of falls | during 6 months
  Fall: an unexpected event in which the participants come to rest on the ground, floor, or lower level.
Safety of interventions | During 6 months
  Pain, headache, itching or soreness on the legs, erythema.

CONTACTS AND LOCATIONS:
Overall Officials: Mercè Sitjà Rabert, PhD, Principal Investigator — • Health Sciences Faculty Blanquerna (Universitat Ramon Llull)
Locations (10):
- Spain (10):
  - Albada Centre Socio Sanitari Parc Taulí, Sabadell, Babadell
  - Ballesol Badalona, Badalona, Barcelona
  - Ballesol Barberà, Barbera Del Valles, Barcelona
  - Residència Poble Nou, Barcelona, Barcelona
  - Ballesol Fabra i Puig, Barcelona, Barcelona
  - Ballesol Almogàvers, Barcelona, Barcelona
  - Residència Mapfre Quavitae, Barcelona, Barcelona
  - Residència AMMA Horta, Barcelona, Barcelona
  - Residència Collserola (Mutuam), Barcelona, Barcelona
  - Residència Allegra, Sabadell, Barcelona

REFERENCES:
- [Derived] Sitja-Rabert M, Martinez-Zapata MJ, Fort Vanmeerhaeghe A, Rey Abella F, Romero-Rodriguez D, Bonfill X. Effects of a whole body vibration (WBV) exercise intervention for institutionalized older people: a randomized, multicentre, parallel, clinical trial. J Am Med Dir Assoc. 2015 Feb;16(2):125-31. doi: 10.1016/j.jamda.2014.07.018. Epub 2014 Oct 3. PMID 25282631
- [Derived] Sitja-Rabert M, Martinez-Zapata MJ, Fort-Vanmeerhaeghe A, Rey-Abella F, Romero-Rodriguez D, Bonfill X. Whole body vibration for older persons: an open randomized, multicentre, parallel, clinical trial. BMC Geriatr. 2011 Dec 22;11:89. doi: 10.1186/1471-2318-11-89. PMID 22192313